CLINICAL TRIAL: NCT06157931
Title: Resilient Students Training (ReST): A Pilot Randomized Controlled Trial
Brief Title: Resilient Students Training (ReST) : A Pilot RCT
Acronym: ReST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, HO Wing Ka Grace, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSEARS20230815002_1
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Psychological Wellness
Keywords: Resilience; Mental Health; University Students; Resilient Student Training Intervention; Adverse Childhood Experiences; Depression; Anxiety; Stress
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Open label parallel-group pilot RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilient Student Training intervention (ReST) (Experimental): Each participant will receive 3 intervention sessions over a 6-week period (1 individual 60-minute session and two 90-minute group-based sessions) delivered by the same interventionist. The specific skills, intervention protocol and intervention manual will be developed in the Phase 1. The skills and exercises will aim to address pertinent areas of needs relating to self-concept, emotional awareness, and maintaining relationships. The individual session will be conducted based on self-assessment results, identifying presenting concerns and goal planning. Group sessions will be gamified to enhance engagement and reward progress. The first group session will build on the individual session's content in a group setting, with the aim to learn from peers. The second group session aims to reinforce the principles and skills learned in the individual session and group session 1 and plan for the future.
  Interventions: Behavioral: Resilient Student Training intervention (ReST)
- Waitlist Control (No Intervention): The waitlist control group will not receive any additional support or interventions whilst waiting to receive the ReST intervention. These participants will be asked to report any psychological interventions or psychotropic medications that they have accessed outside of the trial whilst they are on the waiting list. Wait list control participants will be offered the ReST intervention following their 6-week follow-up assessment.

INTERVENTIONS:
Behavioral: Resilient Student Training intervention (ReST) — ReST consists of one individual 60-minute session and two 90-minute group-based sessions.
  Arms: Resilient Student Training intervention (ReST)

SUMMARY:
Resilience is the ability to survive and thrive despite significant adversity. Trials of resilience-promoting interventions for university students have shown significant improvements in students' resilience and reductions in depressive and stress symptoms. Therefore, the goal of this study is to examine the feasibility of Resilient Student Training Intervention (ReST) to enhance resilience and reduce symptoms of depression, anxiety, and stress in university students with at least one adverse childhood experience (ACE) in Hong Kong.

The study will be conducted in two phases. Phase 1 is a co-designing approach with local university students to discover, define, develop, and deliver the ReST intervention based on the Double Diamond model (Design Council, 2015). In Phase 2, eligible participants will be randomly allocated to either receive the ReST intervention or a waitlist control group. In the intervention group, participants will receive one 60-minute individual session and two 90-minute group-based sessions.

Our main objectives in this study are to answer the following research questions:

1. Can an effective Resilience Student Training Intervention (ReST) be used to improve resilience among undergraduate students with adverse childhood experiences and mental distress?
2. What proportion of eligible individuals participate, engage, and complete the interventions as part of the trial?
3. What proportion of eligible individuals participate in, engage with, and complete research assessments, and what data quality and completion rates can therefore be obtained?
4. Is the ReST intervention safe and acceptable from the participants' perspectives?
5. What sample size is required for a definitive trial?

DETAILED DESCRIPTION:
INTRODUCTION

The occurrence of childhood adversities is more common than previously thought. A recent survey showed that 62% of Hong Kong adults have at least one adverse childhood experience (ACE; a serious, potentially traumatic, and life-altering stressor that occurs before age 18), and nearly 40% have 2 or more ACEs. Resilience was not only protective of mental health but a stronger predictor of mental health status than their ACE history. Existing resilience-promoting interventions for university students have shown improvements in their well-being, but only with small effect sizes and overall low quality of evidence; most trials also involve well-functioning students with unknown trauma histories. Further, existing interventions include a broad spectrum of intervention strategies informed by a wide range of individual and systemic resilience-promoting factors, but all interventions tested to date used a one-size-fits-all approach to improve student resilience without addressing underlying differences in how the resilience process manifests for different individuals. In response, the Youth Resilience Process Model was developed to explain divergent pathways in the youth resilience process based on typologies of initial response to adversity. The model is used to underpin the design of the ReST intervention in this study. In the present study, a Resilient Student Training intervention (ReST) will be co-designed with university students and evaluate the feasibility of a full-scale randomized controlled trial of the intervention. This involves preliminary testing of whether the intervention results in improvements in resilience.

AIMS AND OBJECTIVES

This study aims to (1) Co-design and develop a Resilient Student Training intervention (ReST) so that it can be used with undergraduate students, (2) Test feasibility, acceptability, and safety of the ReST intervention in students with low resilience, adverse childhood experiences, and moderate to severe levels of mental distress, (3) Assess recruitment/retention rates, data quality, and trial procedures for a definitive RCT, and (4) Explore student participants' experiences of taking part in the trial and the intervention to inform subsequent modifications to the intervention and trial design.

METHOD

This study will be conducted in collaboration with a co-designing team comprised of university students who had experience of ACEs, and an experienced multi-disciplinary research team selected based on their clinical, academic, and methodological experience and expertise in all relevant areas. The entire study will be conducted in two phases.

i. PHASE 1

i(a).STUDY DESIGN

A co-designing approach based on the Double Diamond model has been used to "discover", "define", "develop", and "deliver" the ReST intervention. The "discover" stage aims to better understand the problems and support needs of students who have had ACEs and mental distress. The "define" stage uses insights gained from the first stage to define the problem and in the subsequent stage ("develop") brainstorming is used to design, test, and identify appropriate and potentially effective evidence-based typologies-focused therapeutic exercises. The final stage ("deliver") involves pilot testing the exercises on a small scale so that the intervention contents may be improved for use in the subsequent pilot trial. At the point of trial registration (11/2023), co-designing was completed up to the deliver stage. The ReST intervention will consist of one 60-minute individual session and two 90-minute group-based sessions. Each individual session will be adapted to the student's baseline assessment. The first group session will aim to equip students with foundation-level resilience-building skills, which will be built upon during the subsequent advanced skills group sessions. The co-designed interventions will be reported in accordance with the template for intervention description and replication (TIDieR) checklist to ensure the interventions are described in sufficient detail to allow replication.

i(b). PARTICIPANTS AND PROCEDURES

Between 8-16 university students will be recruited by convenience sampling to participate in the pilot study, which constitutes the final "deliver" stage. This single group pre-post pilot study will help the research team establish participants' views on the acceptability and efficacy of the intervention and finalise the intervention contents/exercises. Open-ended questions will be asked to provide their impressions and suggestions in the pilot testing. Data will be collated into themes, and modifications will be made to the intervention or alternative outcome measures will be considered as appropriate.

ii. PHASE 2

ii(a). STUDY DESIGN

This phase will adopt an open-label parallel-group pilot RCT to test the feasibility of ReST to enhance resilience and reduce symptoms of depression, anxiety, and stress in university students with at least one ACE. University student participants will be randomly allocated to either receive the ReST intervention or a waitlist control group. Data collection will be collected at week 0 (baseline), week 6 (post-intervention), and week 10 (follow-up). Each of the three ReST sessions (1 individual session and 2 group-based sessions) is structurally equivalent and will be delivered by the trained interventionists. The intervention will be delivered following a protocol and intervention manual developed in Phase 1. The manual will contain details of all the interventions offered so that all participants have the option to learn coping strategies and skills that are not covered in the sessions as they may find these helpful. The waitlist control group will not receive any additional support or interventions whilst waiting to receive the ReST intervention. These participants will be asked to report any psychological interventions or psychotropic medications that they have accessed outside of the trial whilst they are on the waiting list. Waitlist control participants will be offered the ReST intervention following the completion of their follow-up assessment.

ii(b). PARTICIPANTS AND PROCEDURES

Fifty university student participants will be recruited in each group (ReST intervention and waitlist control), totaling 100 participants. This meets the minimum requirement of 15 participants per arm after 40% attrition. This is also in line with recommendations that feasibility studies of RCTs with two groups should aim for sample sizes of between 24 and 50 participants. An attrition rate of 40% was conservatively assumed as this is a new intervention and no data on drop-out rates was available. All undergraduate students in one local university with (1) at least one ACE (based on the WHO ACE-IQ), (2) low resilience (based on BRS score between 1.00-2.99), and (3) moderate to severe levels of depression, anxiety, or stress (based on DASS-21 cut-offs) will be eligible to participate. Students will complete an online mental health self-assessment and be notified of their eligibility to participate if they meet the above criteria. Exclusion criteria are (1) diagnosis of any mental illness; (2) developmental disability; (3) extremely severe levels of depression, anxiety, or stress (based on DASS-21 cut-offs); and (4) receiving any mental health or psychiatric service or resilience-promoting interventions currently or within the past 6 months. Only adults aged 18 or above who are able to consent to research will be included in the study.

Students will be randomized (1:1) at the start of session 1 to intervention or wait-list control, using randomly permuted block sizes (block sizes of two or four), administered via sealed envelope (an external trial randomization service). Once eligible students have provided their informed consent and completed baseline measures, they will be allocated a unique participant ID number. The trial coordinator will input this ID number into the sealed envelope online system and be immediately informed via email which group the student is randomly allocated to. The internal validity of the trial is strengthened using the external randomization service as the allocation sequence remains concealed because it is retained by the service.

ii(c). OUTCOME MEASURES

Outcomes include retention and data completion rates at each data collection timepoint (baseline, post-intervention, and follow-up) on measures of resilience (BRS; primary outcome), depression, anxiety, and stress (DASS-21; secondary outcome); posttraumatic stress symptoms (ITQ; secondary outcome); adverse events; and 6-month recruitment rate. Baseline information on demographics and ACEs will be gathered to characterize the sample. All study participants will be asked to provide written qualitative feedback on their experiences of taking part in the trial, specifically their views on what worked; what did not work; what could be done differently; and what could be improved. A sample of 12 participants allocated to the intervention condition will be purposively selected (two from each response typology, two that fully completed the trial, and two that withdrew after one intervention session) to participate in individual semi-structured interviews. The interviews will focus on their experiences of engaging in the intervention and participating in the study more broadly.

ii(d). DATA ANALYSIS

Blind analysis of outcome data will be conducted. Proportions, means, SDs, effect sizes, and 95% CIs for all time points will be reported descriptively, on both a strict intention-to-treat and per-protocol basis (>50% attendance in intervention and wait-list control). Missing data due to attrition will be minimized by late randomization (start of intervention session 1) and two phone contacts with participants between assessments. Generalized estimating equation (GEE) will be used for preliminary analysis of intervention efficacy. The intention-to-treat principle dictates that all participants randomized to a treatment condition will be analyzed irrespective of withdrawal. GEE can account for outcome data missing completely at random and where other analysis approaches (i.e., multiple imputations) will be used for any missing data. Interview data will be analyzed via an inductive thematic analysis procedure that follows Braun and Clarke's thematic analysis procedure. Initially, the researchers will immerse themselves in the data set, use line-by-line coding to identify preliminary codes, and develop initial themes. The researchers will then discuss the initial themes and revise them accordingly to define and describe the final themes.

ETHICAL CONSIDERATIONS

Approval has been obtained from the University (HSEARS20230815002). Given that the study participants are students at the university where the study is being conducted there is a potential power imbalance and resulting risk that potential participants may feel coerced to take part. To minimize this risk, participants will be recruited by a Research Assistant that has no role or responsibilities in the students' academic studies. The research team will strictly follow the Good Clinical Practice guidelines for recording, coding, and managing adverse events. All adverse events that occur during the trial will be reported to the principal investigator immediately and to the trial steering committee within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Current PolyU undergraduate student;
2. Low resilience (based on the BRS score between 1.00-2.99);
3. Moderate to severe depression, anxiety, or stress (based on the DASS-21 cut-offs); and
4. Self-report of at least one ACE (based on the WHO ACE-IQ).

Exclusion Criteria:

1. Diagnosis of any mental illnesses;
2. Developmental disability;
3. Extremely severe levels of depression, anxiety, or stress (based on DASS-21 cut-offs); and
4. Receiving any mental health or psychiatric service or resilience-promoting interventions currently or within the past 6 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Week 0 (baseline), Week 6 (post-intervention), and Week 10 (follow-up).
  Proportion of eligible individuals who consent, participate, and complete the intervention/ research assessments.
Acceptability of the intervention | Week 6 (post-intervention) and Week 10 (follow-up).
  Quantitative measure of participant satisfaction based on a 5-point Likert scale ranging from "1=Very Dissatisfied" to "5=Very Satisfied," and qualitative description of participants' perspectives on acceptability of the intervention.
Safety of the intervention based on number of adverse events | Week 0 (baseline), Week 6 (post-intervention), and Week 10 (follow-up).
  Number and type of adverse events will be recorded.
Resilience | Week 0 (baseline), Week 6 (post-intervention), and Week 10 (follow-up).
  The Brief Resilience Scale (BRS), a 6-item self-report questionnaire that measures perceived ability to bounce back from adversity will be used. Responses are provided on a 5-point Likert scale ranging from "strongly disagree=1" to "strongly agree=5." Scores are calculated based on the average of the 6 items, with cut-offs defined as low resilience (1-2.99), normal (3-4.30), and high (4.31-5.0). The Chinese BRS demonstrated good internal consistency, criterion validity, and construct validity when applied in university undergraduate students (Fung, 2020).

SECONDARY OUTCOMES:
Depression | Week 0 (baseline), Week 6 (post-intervention), and Week 10 (follow-up).
  The Depression, Anxiety, Stress Scale (DASS-21) is a well-validated tool commonly used to measure psychological distress (Oei et al., 2013). The self-completed measure consists of seven questions for each of the three subscales (Depression, Anxiety and Stress). Each question is scored on a four-point Likert scale (0=never, 1=sometimes, 2=often and 3=almost always). The DASS-12 is reported to have sound psychometric properties in a wide range of clinical and non-clinical populations, including good internal consistency and concurrent validity with the original DASS-42 (Antony et al., 1998).
Anxiety | Week 0 (baseline), Week 6 (post-intervention), and Week 10 (follow-up).
  The Depression, Anxiety, Stress Scale (DASS-21) is a well-validated tool commonly used to measure psychological distress (Oei et al., 2013). The self-completed measure consists of seven questions for each of the three subscales (Depression, Anxiety and Stress). Each question is scored on a four-point Likert scale (0=never, 1=sometimes, 2=often and 3=almost always). The DASS-12 is reported to have sound psychometric properties in a wide range of clinical and non-clinical populations, including good internal consistency and concurrent validity with the original DASS-42 (Antony et al., 1998).
Stress | Week 0 (baseline), Week 6 (post-intervention), and Week 10 (follow-up).
  The Depression, Anxiety, Stress Scale (DASS-21) is a well-validated tool commonly used to measure psychological distress (Oei et al., 2013). The self-completed measure consists of seven questions for each of the three subscales (Depression, Anxiety and Stress). Each question is scored on a four-point Likert scale (0=never, 1=sometimes, 2=often and 3=almost always). The DASS-12 is reported to have sound psychometric properties in a wide range of clinical and non-clinical populations, including good internal consistency and concurrent validity with the original DASS-42 (Antony et al., 1998).
Posttraumatic Stress | Week 0 (baseline), Week 6 (post-intervention), and Week 10 (follow-up).
  International Trauma Questionnaire (ITQ) will be used to assess symptoms of ICD-11 PTSD and CPTSD. Six questions measure the PTSD symptoms (re-experiencing, avoidance, sense of current threat) and six questions measure the DSO symptoms (affective dysregulation, negative self-concept, and disturbed relationships). Three additional items measure functional impairment. The measure has been shown to have good psychometric properties when used with Hong Kong University students (Ho, Karatzias, et al., 2019).

OTHER OUTCOMES:
Experiences of the intervention/trial | Week 6 (post-intervention), and Week 10 (follow-up).
  Study participants will provide written qualitative feedback on their experiences of taking part in the trial, specifically their views on what worked; what did not work; what could be done differently; and what could be improved. Semi-structured interviews will be conducted to extract their experiences of engaging in the intervention and participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Grace WK Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, Hong Kong, Hong Kong

REFERENCES:
- [Background] Ang WHD, Lau ST, Chen, LJ, Chew HSJ, Tan JH, Shorey S, Lau Y. Effectiveness of resilience interventions for higher education students: A meta-analysis and metaregression. J Educ Psychol. 2022 Oct;114(7):1670-94. doi: 10.1037/edu0000719
- [Background] Design Council. The Double Diamond: A universally accepted depiction of the design process. Retrieved May 17, 2023 from https://www.designcouncil.org.uk/our-resources/the-double- diamond/
- [Background] Dube SR, Anda RF, Felitti VJ, Chapman DP, Williamson DF, Giles WH. Childhood abuse, household dysfunction, and the risk of attempted suicide throughout the life span: findings from the Adverse Childhood Experiences Study. JAMA. 2001 Dec 26;286(24):3089-96. doi: 10.1001/jama.286.24.3089. PMID 11754674
- [Background] Fung SF. Validity of the Brief Resilience Scale and Brief Resilient Coping Scale in a Chinese Sample. Int J Environ Res Public Health. 2020 Feb 16;17(4):1265. doi: 10.3390/ijerph17041265. PMID 32079115
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Ho GWK, Chan ACY, Chien WT, Bressington DT, Karatzias T. Examining patterns of adversity in Chinese young adults using the Adverse Childhood Experiences-International Questionnaire (ACE-IQ). Child Abuse Negl. 2019 Feb;88:179-188. doi: 10.1016/j.chiabu.2018.11.009. Epub 2018 Dec 2. PMID 30513406
- [Background] Ho GWK, Chan ACY, Shevlin M, Karatzias T, Chan PS, Leung D. Childhood Adversity, Resilience, and Mental Health: A Sequential Mixed-Methods Study of Chinese Young Adults. J Interpers Violence. 2021 Oct;36(19-20):NP10345-NP10370. doi: 10.1177/0886260519876034. Epub 2019 Sep 15. PMID 31524036
- [Background] Ho GWK, Karatzias T, Cloitre M, Chan ACY, Bressington D, Chien WT, Hyland P, Shevlin M. Translation and validation of the Chinese ICD-11 International Trauma Questionnaire (ITQ) for the Assessment of Posttraumatic Stress Disorder (PTSD) and Complex PTSD (CPTSD). Eur J Psychotraumatol. 2019 May 15;10(1):1608718. doi: 10.1080/20008198.2019.1608718. eCollection 2019. PMID 31143410
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Oei TP, Sawang S, Goh YW, Mukhtar F. Using the Depression Anxiety Stress Scale 21 (DASS-21) across cultures. Int J Psychol. 2013;48(6):1018-29. doi: 10.1080/00207594.2012.755535. Epub 2013 Feb 21. PMID 23425257
- [Background] Antony MM, Bieling PJ, Cox BJ, Enns MW, Swinson RP. Psychometric Properties of the 42-item and 21-item versions of the depression anxiety stress scales in clinical groups and a community sample. Psychol Assess. 1998;10(2): 176-81. doi:10.1037/1040-3590.10.2.176.